CLINICAL TRIAL: NCT04876196
Title: Evaluation of a 12-Week Web-Based Intervention for Bulimia Nervosa: a Randomized Controlled Trial
Brief Title: Evaluation of a Web-Based Intervention for Bulimia Nervosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: Selfapy GmbH (Unknown)
Responsible Party: Principal Investigator, Christina Timm, Principal Investigator, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Selfapy-BN
Record Dates: First submitted 2021-05-02; First posted 2021-05-06 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Bulimia Nervosa
Keywords: Ecological Momentary Assessment; Internet-based Intervention; Randomized Controlled Trial
MeSH Terms: conditions — Bulimia Nervosa

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with an intervention group and a waiting list control group
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants are blinded about the two conditions of the study and told that the assigned waiting time for the web-based intervention varies randomly. Therefore, participants in the control group do not know that the other group starts the intervention immediately. However, complete masking of participants is precluded as all subjects are aware of when they get access to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Active Comparator): Web-based intervention (Selfapy for Bulimia Nervosa)
  Interventions: Other: Selfapy for Bulimia Nervosa
- Waitlist Control Group (No Intervention): 12-week waiting period

INTERVENTIONS:
Other: Selfapy for Bulimia Nervosa — Web-based intervention for Bulimia Nervosa with six mandatory weekly sessions covering topics related to eating behaviors, emotion regulation, and stress management, followed by an optional set of up to six modular specialization areas based on individual therapy goals. During the intervention, participants can access an online chat providing crisis management, answering questions concerning the exercises, and technical support. The chat does not include the opportunity to discuss individual topics and concerns about treatment.
  Arms: Intervention Group

SUMMARY:
This study evaluates the effectiveness of a web-based intervention specifically designed for patients with Bulimia Nervosa (BN) in a blinded randomized controlled trial.

After a sign-up process, a diagnostic interview, and a baseline assessment, eligible participants will be randomly allocated either to (1) an intervention group including the online web-based intervention for BN or (2) a waitlist control group with delayed access to the intervention (12 weeks). The program comprises six mandatory weekly sessions and six modular specialization areas resulting in a treatment period of 12 weeks. Minimal guidance is provided via a chat function.

Assessments will be conducted at pretreatment (study entrance), six weeks after baseline (mid-treatment), and 12 weeks after baseline (post-treatment).

The investigators expect that the intervention group will show lower frequencies of binge eating episodes and compensatory behavior as the primary outcome variables after the 12 weeks of treatment compared to a waitlist control condition. Moreoever, the investigators assume that there will be a higher reduction in global eating disorder symptoms, comorbid psychopathology, and a higher increase in well-being and self-esteem over 12 weeks in the intervention group compared to the waitlist control group.

Finally, the investigators expect that the intervention group will demonstrate a significantly higher reduction in functional impairment, substantially better restoration of work capacity, and an improved ability to regulate emotions after the 12 weeks of treatment.

DETAILED DESCRIPTION:
Background: Bulimia Nervosa (BN) is characterized by persistent episodes of uncontrolled eating and inappropriate compensatory behaviors, associated with marked impairments in physical and mental health, social integration, professional performance, and overall quality of life. Although cognitive-behavioral therapies are effective for bulimia nervosa, access to specialized treatment in Germany is limited due to patient-related barriers and insufficient healthcare resources. Internet-based interventions can overcome this treatment gap and reduce the burden of BN for both patients and the healthcare system by making evidence-based interventions more accessible.

Goal: This study evaluates the effectiveness of a web-based intervention specifically designed for patients with BN in a blinded randomized controlled trial.

Method: After a sign-up process, a structured diagnostic interview, and a baseline assessment, eligible participants will be randomly allocated either to (1) an intervention group including the online web-based intervention for BN or (2) a waitlist control group with delayed access to the intervention (12 weeks). The program comprises six mandatory weekly sessions covering topics related to eating behaviors, emotion regulation, and stress management, followed by an optional set of up to six modular specialization areas based on individual therapy goals. Moreover, minimal guidance is included, consisting of technical support and answering questions via a chat function. Assessments will be conducted at pretreatment (study entrance), six weeks after baseline (mid-treatment), and 12 weeks after baseline (post-treatment). The primary outcome will be the number of binge eating episodes and compensatory behaviors. Secondary measures include global eating pathology, comorbid psychopathology, quality of life, self-esteem, emotion regulation, work capacity, and functional impairments.

Statistical Analyses: An intention-to-treat analysis will be performed to examine differences between the intervention and the control group in the change of eating disorder symptoms and secondary outcomes from pre- to post-treatment.

Hypotheses: The investigators expect that the intervention group will show lower frequencies of binge eating episodes and compensatory behavior as the primary outcome variables after the 12 weeks of treatment compared to a waitlist control condition. The investigators assume that there will be a higher reduction in global eating disorder symptoms, comorbid psychopathology, and a higher increase in well-being and self-esteem over 12 weeks in the intervention group compared to the waitlist control group. Moreover, the investigators expect that the intervention group will demonstrate a significantly higher reduction in functional impairment, substantially better restoration of work capacity, and an improved ability to regulate negative emotions after the 12 weeks of treatment.

ELIGIBILITY:
Inclusion criteria:

* sufficient German language skills (C1)
* permanent internet access during the study period
* meeting the diagnostic criteria for Bulimia Nervosa according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-5)

Exclusion criteria:

* current severe depressive episode
* acute suicidality
* comorbid bipolar disorder or psychotic disorders
* acute substance dependence
* current psychotherapy or pharmacotherapy for eating disorders
* Body Mass Index (BMI) below 18.5

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-07-07 (Actual)

PRIMARY OUTCOMES:
Changes in the frequency of binge eating episodes and compensatory behavior within the last 28 days | 0 weeks, 6 weeks, 12 weeks
  The Eating Disorders Examination Questionnaire (EDE-Q; Berg et al., 2012) captures the frequency of binge eating episodes and compensatory behavior within the last 28 days using 6 items. Higher values indicate a higher frequency of relevant eating disorder episodes.

SECONDARY OUTCOMES:
Changes in global eating psychopathology | 0 weeks, 6 weeks, 12 weeks
  The Eating Disorders Examination Questionnaire (EDE-Q; Berg et al., 2012) allows assessing global eating psychopathology based on 22 items. Mean scores range from 0 to 6, with higher values indicating a higher global eating psychopathology.
Changes in the weekly frequency of binge eating episodes, compensatory behavior, and regular eating | 0 weeks, 1 week, 2 weeks, 3 weeks, 4 weeks, 5 weeks, 6 weeks, 7 weeks, 8 weeks, 9 weeks, 10 weeks, 11 weeks, 12 weeks
  The Weekly Binges Questionnaire (WBQ; Munsch et al., 2007) assesses the frequency of binge eating episodes, compensatory behavior, and regular eating by asking participants to count the number of binge eating episodes, the number of compensatory behaviors, and the number of days with regular eating habits. While a higher number of binges and compensatory behaviors indicates a higher symptomatology, a higher number of regular eating days indicates a lower symptomatology.
Changes in everyday eating disorder symptoms | 0 weeks, 12 weeks
  Ecological momentary assessment (EMA) of eating disorder symptoms (shape concerns, weight concerns, binge eating episodes, episodes of compensatory behaviors, urges to eat or compensate) for five days (five signal-contingent measurements and additional event-contingent assessments)
Changes in eating-disorder-related daily difficulties | 0 weeks, 6 weeks, 12 weeks
  The Clinical Impairment Assessment Questionnaire (CIA; Bohn et al., 2008) consists of 16 items answered on a 4-point Likert scale. The overall score ranges from 0 to 48. Higher values indicate a higher level of clinical impairment.
Changes in comorbid depressive symptoms | 0 weeks, 6 weeks, 12 weeks
  The Patient Health Questionnaire (PHQ-9; Kroenke et al., 2001) consists of 9 items answered on a 4-point scale. The overall score ranges from 0 to 27. Higher values indicate a higher level of depressive symptomology.
Changes in comorbid anxiety symptoms | 0 weeks, 6 weeks, 12 weeks
  The General Anxiety Disorder Scale (GAD-7; Spitzer et al., 2006) consists of 7 items answered on a 4-point scale. The overall score ranges from 0 to 21. Higher values indicate a higher level of anxiety symptoms.
Changes in well-being | 0 weeks, 6 weeks, 12 weeks
  The World Health Organization Well-Being Index (WHO-5; Topp et al., 2015) consists of 5 items answered on a 6-point scale. The overall score ranges from 0 to 100. Higher values indicate a higher level of well-being.
Changes in self-esteem | 0 weeks, 6 weeks, 12 weeks
  The Rosenberg Self-Esteem Scale (RSES; Roth et al., 2008) consists of 10 items answered on a 4-point scale. The overall score ranges from 0 to 30. Higher values indicate a higher level of self-esteem.
Changes in work capacity | 0 weeks, 6 weeks, 12 weeks
  The iMTA Productivity Cost Questionnaire (iPCQ; Bouwmans et al., 2015) consists of 12 items grouped in general questions about paid work and questions about productivity losses in paid and unpaid work. The questionnaire captures the missed work time (paid and unpaid) in hours for short-term absence and calendar days for long-time absence and the hours of lost productivity due to presenteeism.
Changes in emotion regulation frequencies | 0 weeks, 6 weeks, 12 weeks
  The Heidelberg Form for Emotion Regulation Strategies (HFERST; Izadpanah et al., 2019) consists of 28 items answered on a 5-point scale. For each of the eight emotion regulation strategies (rumination, reappraisal, acceptance, problem solving, suppression of emotional expression, suppression of emotional experience, avoidance, social support), a score ranging from 1 to 5 can be calculated. Higher values indicate a higher frequency of emotion regulation strategy endorsement.
Changes in emotion regulation difficulties | 0 weeks, 6 weeks, 12 weeks
  The Difficulties in Emotion Regulation Scale (DERS; Gratz & Roemer, 2004) consists of 36 items answered on a 5-point scale. The overall score ranges from 36 to 180. Higher values indicate a higher level of emotion regulation difficulties.
Changes in everyday emotion regulation | 0 weeks, 12 weeks
  Ecological momentary assessment (EMA) of affect, emotion regulation strategies and difficulties for five days (five signal-contingent measurements, and additional event-contingent assessments)

OTHER OUTCOMES:
Changes in attitudes towards psychological online interventions | 0 weeks, 12 weeks
  Two subscales of the Attitudes Towards Psychological Online Interventions Scale (APOI; Schroeder et al., 2015) will be used. These capture technologization threat and perceived anonymity benefits using 8 items on a 5-point scale. Higher values indicate a more positive attitude towards psychological online interventions.
Changes in patient outcome expectancies | 0 weeks, 6 weeks (intervention group), 12 weeks
  The Patients' Therapy Expectation and Evaluation Scale (PATHEV; Schulte, 2008) consists of 16 items answered on a 5-point scale. The overall score ranges from 0 to 5. Higher values indicate more positive expectancies towards the therapy.
Negative intervention effects | 6 weeks (intervention group), 12 weeks
  The Negative Effects Questionnaire (NEQ; Rozental et al., 2019) consists of 32 items. For each item, the participants answer whether the adverse effect occurred (yes/no), how strong the negative effect was (0 to 4) and whether they attribute the negative effect on the treatment or something else. Two scores can be obtained, one for the frequency of adverse effects due to treatment, ranging from 0 to 32, and one for the negative impact, ranging from 0 to 128. Higher values indicate a higher level of adverse effects.
Use of other healthcare services | 0 weeks, 6 weeks, 12 weeks
  The Client Sociodemographic Service Receipt Inventory - European Version (CSSRI-EU; Chisholm et al., 2000) allows assessing the number and length of using different types of healthcare services. Higher values indicate a higher number and frequency of healthcare service usage.

CONTACTS AND LOCATIONS:
Overall Officials: Luise Pruessner, Principal Investigator — Department of Psychology, Heidelberg University; Christina Timm, PhD, Principal Investigator — Department of Psychology, Heidelberg University; Steffen Hartmann, Principal Investigator — Department of Psychology, Heidelberg University; Sven Barnow, Prof., Principal Investigator — Department of Psychology, Heidelberg University
Locations (1):
- Heidelberg University, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be uploaded after publication of the results.

REFERENCES:
- [Background] Berg KC, Peterson CB, Frazier P, Crow SJ. Psychometric evaluation of the eating disorder examination and eating disorder examination-questionnaire: a systematic review of the literature. Int J Eat Disord. 2012 Apr;45(3):428-38. doi: 10.1002/eat.20931. Epub 2011 Jul 8. PMID 21744375
- [Background] Bohn K, Doll HA, Cooper Z, O'Connor M, Palmer RL, Fairburn CG. The measurement of impairment due to eating disorder psychopathology. Behav Res Ther. 2008 Oct;46(10):1105-10. doi: 10.1016/j.brat.2008.06.012. Epub 2008 Jul 2. PMID 18710699
- [Background] Bouwmans C, Krol M, Severens H, Koopmanschap M, Brouwer W, Hakkaart-van Roijen L. The iMTA Productivity Cost Questionnaire: A Standardized Instrument for Measuring and Valuing Health-Related Productivity Losses. Value Health. 2015 Sep;18(6):753-8. doi: 10.1016/j.jval.2015.05.009. Epub 2015 Aug 20. PMID 26409601
- [Background] Chisholm D, Knapp MR, Knudsen HC, Amaddeo F, Gaite L, van Wijngaarden B. Client Socio-Demographic and Service Receipt Inventory--European Version: development of an instrument for international research. EPSILON Study 5. European Psychiatric Services: Inputs Linked to Outcome Domains and Needs. Br J Psychiatry Suppl. 2000;(39):s28-33. doi: 10.1192/bjp.177.39.s28. PMID 10945075
- [Background] Gratz, K. L., & Roemer, L. (2004). Multidimensional assessment of emotion regulation and dysregulation: Development, factor structure, and initial validation of the difficulties in emotion regulation scale. Journal of psychopathology and behavioral assessment, 26(1), 41-54.
- [Background] Izadpanah S, Barnow S, Neubauer AB, Holl J. Development and Validation of the Heidelberg Form for Emotion Regulation Strategies (HFERST): Factor Structure, Reliability, and Validity. Assessment. 2019 Jul;26(5):880-906. doi: 10.1177/1073191117720283. Epub 2017 Jul 21. PMID 28730850
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Munsch S, Biedert E, Meyer A, Michael T, Schlup B, Tuch A, Margraf J. A randomized comparison of cognitive behavioral therapy and behavioral weight loss treatment for overweight individuals with binge eating disorder. Int J Eat Disord. 2007 Mar;40(2):102-13. doi: 10.1002/eat.20350. PMID 17089420
- [Background] Roth, M., Decker, O., Herzberg, P. Y., & Brähler, E. (2008). Dimensionality and norms of the Rosenberg Self-Esteem Scale in a German general population sample. European Journal of Psychological Assessment, 24(3), 190-197.
- [Background] Rozental A, Kottorp A, Forsstrom D, Mansson K, Boettcher J, Andersson G, Furmark T, Carlbring P. The Negative Effects Questionnaire: psychometric properties of an instrument for assessing negative effects in psychological treatments. Behav Cogn Psychother. 2019 Sep;47(5):559-572. doi: 10.1017/S1352465819000018. Epub 2019 Mar 15. PMID 30871650
- [Background] Schroder J, Sautier L, Kriston L, Berger T, Meyer B, Spath C, Kother U, Nestoriuc Y, Klein JP, Moritz S. Development of a questionnaire measuring Attitudes towards Psychological Online Interventions-the APOI. J Affect Disord. 2015 Nov 15;187:136-41. doi: 10.1016/j.jad.2015.08.044. Epub 2015 Aug 28. PMID 26331687
- [Background] Schulte D. Patients' outcome expectancies and their impression of suitability as predictors of treatment outcome. Psychother Res. 2008 Jul;18(4):481-94. doi: 10.1080/10503300801932505. PMID 18815999
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Topp CW, Ostergaard SD, Sondergaard S, Bech P. The WHO-5 Well-Being Index: a systematic review of the literature. Psychother Psychosom. 2015;84(3):167-76. doi: 10.1159/000376585. Epub 2015 Mar 28. PMID 25831962
- [Background] Chih CP, He J, Sly TS, Roberts EL Jr. Comparison of glucose and lactate as substrates during NMDA-induced activation of hippocampal slices. Brain Res. 2001 Mar 2;893(1-2):143-54. doi: 10.1016/s0006-8993(00)03306-0. PMID 11223002
- [Derived] Hartmann S, Timm C, Barnow S, Rubel JA, Lalk C, Pruessner L. Web-Based Cognitive Behavioral Treatment for Bulimia Nervosa: A Randomized Clinical Trial. JAMA Netw Open. 2024 Jul 1;7(7):e2419019. doi: 10.1001/jamanetworkopen.2024.19019. PMID 38958978
- [Derived] Hartmann S, Pruessner L, Rubel JA, Lalk C, Barnow S, Timm C. Applying a web-based self-help intervention for bulimia nervosa in routine care: Study protocol for a randomized controlled trial. Internet Interv. 2022 Feb 17;28:100512. doi: 10.1016/j.invent.2022.100512. eCollection 2022 Apr. PMID 35251938